CLINICAL TRIAL: NCT06967428
Title: Effectiveness of Metabolic Modulation in Treating Post-vaccination Syndrome: A Prospective Study
Brief Title: Effect of Metabolic Modulation on a Post-acute COVID-19 Vaccination Syndrome (PACVS) Cohort
Acronym: ViTAL-SCAN19
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Independent Medical Alliance (Other)
Collaborators: Open Source Medicine Foundation OU (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ViTAL-SCAN for PACVS
Record Dates: First submitted 2025-05-05; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Vaccine Adverse Reaction; Post Acute Covid-19 Vaccination Syndrome
Keywords: Post Acute Covid-19 Vaccination Syndrome; Metabolic Modulation; Amino Acids
MeSH Terms: interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ViTAL SCAN (Experimental): This daily intervention over 3 months combines 4 g L-serine, 14 g L-glutamine, 3 g L-arginine, 2.5 g N-acetylcysteine, 5.75 g L-citrulline, 1 g vitamin C, and 5 g creatine to modulate energy metabolism.
  Interventions: Combination Product: Combined metabolic modulator
- Rice Protein Powder and Vitamin C (Active Comparator): A mass-matched supplement of rice protein powder with vitamin C.
  Interventions: Dietary Supplement: Rice Protein Powder with Vitamin C

INTERVENTIONS:
Combination Product: Combined metabolic modulator — This daily intervention over 3 months combines 4 g L-serine, 14 g L-glutamine, 3 g L-arginine, 2.5 g N-acetylcysteine, 5.75 g L-citrulline, 1 g vitamin C, and 5 g creatine to support energy metabolism.
  Arms: ViTAL SCAN
Dietary Supplement: Rice Protein Powder with Vitamin C — Rice Protein Powder (39g) with Vitamin C (1g) daily
  Arms: Rice Protein Powder and Vitamin C

SUMMARY:
The goal of this clinical trial is to evaluate whether metabolic modulation with a combined nutraceutical product can improve symptoms and metabolic health in adults diagnosed with post-acute Covid-19 vaccination syndrome (PACVS), a condition characterized by persistent fatigue and exercise intolerance attributed to Covid-19 vaccination and confirmed by laboratory testing.

The main questions it aims to answer are:

Does the combined nutraceutical intervention improve quality of life (measured by the PAC-19QoL questionnaire) in PACVS patients?

Does the intervention improve metabolic, inflammatory, and functional biomarkers (e.g., HbA1c, blood lactate, CRP, spike protein levels, heart rate variability, 6-minute walk distance)?

Researchers will compare the intervention group (receiving the ViTAL SCAN nutraceutical) to a placebo group (receiving rice protein powder with vitamin C) to determine if the intervention leads to greater improvements in symptoms and biomarker profiles.

Participants will:

Take the assigned supplement daily for 3 months (ViTAL SCAN or placebo)

Attend clinic visits for blood and urine sampling, physical performance tests (6-minute walk test), and heart rate monitoring

Complete quality of life and health behavior questionnaires

Undergo measurements of metabolic and inflammatory markers (HbA1c, lactate, CRP, spike protein)

Record supplement intake

This study is currently pending IRB approval and aims to enroll 100 adults with PACVS for a randomized, placebo-controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Persistent fatigue lasting more than 6 months
* Received at least one dose of a Covid-19 vaccine, after which they experienced fatigue symptoms (symptom onset within two weeks of vaccination)
* Laboratory result showing persistent spike protein in blood OR presence of spike protein antibodies with SARS-CoV-2 nucleocapsid antibodies negative.

Exclusion Criteria:

* Pregnant
* History of Schizophrenia
* Currently using antidepressant medication

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
PAC-19QoL Questionnaire | From enrollment to an interim measurement at 1.5 months to the end of treatment at 3 months"
  Combined score of an established survey instrument for Quality of Life in the context of Post-Acute Covid-19 Syndrome (PACS).
Six-minute walk test | From enrollment to an interim measurement at 1.5 months to the end of treatment at 3 months"
  A treadmill-administered version of the six minute walk test (6MWT) where patients walk for as long a distance as they can, without jogging or running, in 6 minutes.

SECONDARY OUTCOMES:
Hemoglobin A1c | From enrollment to an interim measurement at 1.5 months to the end of treatment at 3 months"
  Hemoglobin A1c (HbA1c) reflects longer term blood sugar levels. Given that metabolism is altered in PACS patients, it may be valuable to assess their metabolic health. Elevated HbA1c was associated with an increased mortality during the acute phase of the Covid-19.
Sedentary blood lactate | From enrollment to an interim measurement at 1.5 months to the end of treatment at 3 months"
  Blood lactate when the patient is at rest is taken using the Arkray Lactate Pro 2 Sports Blood Lactate Meter, which uses disposable test strips.
Post-exertion blood lactate | From enrollment to an interim measurement at 1.5 months to the end of treatment at 3 months"
  Blood lactate taken after the six-minute walk test.
C-Reactive Protein | From enrollment to an interim measurement at 1.5 months to the end of treatment at 3 months"
  C-reactive protein (CRP) , a marker of inflammation, has been found to be significantly different between long covid groups vs healthy individuals, as well as between long covid and recovered individuals.
  CRP is quantitatively measured at a laboratory attached to the study clinic using the Roche Cobas b 101 Blood Analyser using Roche cobas b 101 CRP Test Discs, supplied in packs of 10. Each test required a 12 μL sample of capillary whole blood, obtained via finger prick.
  Upon completion of the assay, CRP concentrations are recorded in mg/L with that patient's identification number. The analytical range is 3.0-400 mg/L; if a test returns an error, the value will be reported as missing.
Spike protein levels | From an initial test at enrollment to another at the end of treatment at 3 months"
  Spike protein tests will be performed using the MSD S-PLEX SARS-CoV-2 Spike Kit using a SECTOR Imager 2400 plate reader.
Resting Heart Rate Variability | From enrollment to an interim measurement at 1.5 months to the end of treatment at 3 months"
  Heart Rate Variability is taken at rest using a Garmin vívosmart® 5.
Heart rate variability during 6MWT | From enrollment to an interim measurement at 1.5 months to the end of treatment at 3 months"
  HRV is taken using a Garmin vívosmart® 5 at the halfway point of the 6 minute walk test.
Resting Heart Rate | From enrollment to an interim measurement at 1.5 months to the end of treatment at 3 months"
  Resting Heart Rate is taken using a Garmin vívosmart® 5.
Heart Rate during 6MWT | From enrollment to an interim measurement at 1.5 months to the end of treatment at 3 months"
  Average heart rate is taken during the last three minutes of the 6MWT
Post-exercise Borg category-ratio 10 scale | From enrollment to an interim measurement at 1.5 months to the end of treatment at 3 months"
  This test is used to assess the level of perceived exertion after the 6MWT by asking participants to rate their exertion on a scale of 1 to 10. This is useful as a measure of exercise intolerance.
Total Cholesterol | From enrollment to an interim measurement at 1.5 months to the end of treatment at 3 months"
HDL-Cholesterol | From enrollment to an interim measurement at 1.5 months to the end of treatment at 3 months"
LDL-Cholesterol | From enrollment to an interim measurement at 1.5 months to the end of treatment at 3 months"
Triglycerides | From enrollment to an interim measurement at 1.5 months to the end of treatment at 3 months"

CONTACTS AND LOCATIONS:
Locations (1):
- Dorrington Medical Associates, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Demographic data (Age, sex and US census category for ethnicity), Baseline, Interim and final measurements of outcome measures.
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- See also: Study protocol — https://preprints.jmir.org/preprint/70342